CLINICAL TRIAL: NCT05467384
Title: Effect of Amlodipine on the Lipid Profile of Newly Diagnosed Hypertensive Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ayub Teaching Hospital (Other)
Collaborators: Khyber Medical University Peshawar (Other)
Responsible Party: Principal Investigator, Shahid ali shah, Assistant Professor, Ayub Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: sashah0002
Record Dates: First submitted 2021-07-16; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Hypercholesterolemia; Hypertension; Cholesterol Deposition
Keywords: Hypercholesterolemia; Hypertension
MeSH Terms: conditions — Hypercholesterolemia; Hypertension | interventions — Amlodipine

STUDY DESIGN:
Intervention Model Description: Case with healthy control
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Newly Diagnosed Hypertensive patients (Experimental): These are the patients that have been clearly diagnosed with diabetes for the first time.
  Interventions: Drug: Amlodipine
- Healthy Controls (No Intervention): Healthy Control Group

INTERVENTIONS:
Drug: Amlodipine — 5mg/day in two divided doses
  Other Names: Norvasc
  Arms: Newly Diagnosed Hypertensive patients

SUMMARY:
In this study, Amlodipine has been used to study its effects in newly diagnosed hypertensive patients.

DETAILED DESCRIPTION:
The incidence of hypertension is on the rise in developing countries like Pakistan. Different medications are used to decrease blood pressure with Amlodipine as one of the first-line drugs. It was proposed that due to interaction with calcium and thus luminal cholecystokinin releasing factor; Amlodipine might increase the cholesterol level and thus cause dyslipidemia.

Objective: In this regard, this study was conducted to look into the effects of Amlodipine in newly diagnosed cases of hypertension that had received no medication previously.

Methodology: Experimental study with a healthy control group with the sample size calculated out to be 80, comprising of an equal number of enrolment into case and control groups.

ELIGIBILITY:
Inclusion criteria for cases.

1) Newly diagnosed mild to moderate hypertensive. (2) Non-obese individuals. 3) Must not have received antihypertensive treatment previously. 4) Has elevated serum cholesterol levels. Exclusion criteria for cases

1) Any other major illness.

Inclusion criteria for controls

1. Normal lipid profile.
2. Normotensive (BP < 140/90mmHg). Exclusion criteria for controls

1) Any major illness.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Measurement of Blood Glucose Concentration | Four Months
  Measured as per protocols provided by the kit manufacturer.
Measurement of Total Plasma Cholesterol Concentration | Four Months
  Measured as per protocols provided by the kit manufacturer.
Measurement of Plasma Triglyceride Concentration | Four Months
  Measured as per protocols provided by the kit manufacturer.
Measurement of Plasma High Density Lipoproteins Concentration | Four Months
  Measured as per protocols provided by the kit manufacturer.
Measurement of Plasma Low Density Lipoproteins Concentration | Four Months
  Measured as per protocols provided by the kit manufacturer.

CONTACTS AND LOCATIONS:
Overall Officials: Shahid A Shah, BDS, MPhil, Principal Investigator — Faculté d'Odontologie, Université de Montpellier

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] James PA, Oparil S, Carter BL, Cushman WC, Dennison-Himmelfarb C, Handler J, Lackland DT, LeFevre ML, MacKenzie TD, Ogedegbe O, Smith SC Jr, Svetkey LP, Taler SJ, Townsend RR, Wright JT Jr, Narva AS, Ortiz E. 2014 evidence-based guideline for the management of high blood pressure in adults: report from the panel members appointed to the Eighth Joint National Committee (JNC 8). JAMA. 2014 Feb 5;311(5):507-20. doi: 10.1001/jama.2013.284427. PMID 24352797
- [Background] Abebe SM, Berhane Y, Worku A, Getachew A. Prevalence and associated factors of hypertension: a crossectional community based study in northwest ethiopia. PLoS One. 2015 Apr 24;10(4):e0125210. doi: 10.1371/journal.pone.0125210. eCollection 2015. PMID 25909382
- [Background] Mancia G, De Backer G, Dominiczak A, Cifkova R, Fagard R, Germano G, Grassi G, Heagerty AM, Kjeldsen SE, Laurent S, Narkiewicz K, Ruilope L, Rynkiewicz A, Schmieder RE, Boudier HA, Zanchetti A, Vahanian A, Camm J, De Caterina R, Dean V, Dickstein K, Filippatos G, Funck-Brentano C, Hellemans I, Kristensen SD, McGregor K, Sechtem U, Silber S, Tendera M, Widimsky P, Zamorano JL, Erdine S, Kiowski W, Agabiti-Rosei E, Ambrosioni E, Lindholm LH, Viigimaa M, Adamopoulos S, Agabiti-Rosei E, Ambrosioni E, Bertomeu V, Clement D, Erdine S, Farsang C, Gaita D, Lip G, Mallion JM, Manolis AJ, Nilsson PM, O'Brien E, Ponikowski P, Redon J, Ruschitzka F, Tamargo J, van Zwieten P, Waeber B, Williams B; Management of Arterial Hypertension of the European Society of Hypertension; European Society of Cardiology. 2007 Guidelines for the Management of Arterial Hypertension: The Task Force for the Management of Arterial Hypertension of the European Society of Hypertension (ESH) and of the European Society of Cardiology (ESC). J Hypertens. 2007 Jun;25(6):1105-87. doi: 10.1097/HJH.0b013e3281fc975a. No abstract available. PMID 17563527
- [Background] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; National Heart, Lung, and Blood Institute Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure; National High Blood Pressure Education Program Coordinating Committee. The Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure: the JNC 7 report. JAMA. 2003 May 21;289(19):2560-72. doi: 10.1001/jama.289.19.2560. Epub 2003 May 14. PMID 12748199
- [Background] Ruilope LM, Burnier M, Muszbek N, Brown RE, Keskinaslan A, Ferber P, Harms G. Public health value of fixed-dose combinations in hypertension. Blood Press Suppl. 2008 Jun;1:5-14. PMID 18705530
- [Background] Saleem F, Hassali AA, Shafie AA. Hypertension in Pakistan: time to take some serious action. Br J Gen Pract. 2010 Jun;60(575):449-50. doi: 10.3399/bjgp10X502182. No abstract available. PMID 20529498
- [Background] Hashmi SK, Afridi MB, Abbas K, Sajwani RA, Saleheen D, Frossard PM, Ishaq M, Ambreen A, Ahmad U. Factors associated with adherence to anti-hypertensive treatment in Pakistan. PLoS One. 2007 Mar 14;2(3):e280. doi: 10.1371/journal.pone.0000280. PMID 17356691
- [Background] Johnson LK, Hofso D, Aasheim ET, Tanbo T, Holven KB, Andersen LF, Roislien J, Hjelmesaeth J. Impact of gender on vitamin D deficiency in morbidly obese patients: a cross-sectional study. Eur J Clin Nutr. 2012 Jan;66(1):83-90. doi: 10.1038/ejcn.2011.140. Epub 2011 Jul 27. PMID 21792214
- [Background] van Ballegooijen AJ, Cepelis A, Visser M, Brouwer IA, van Schoor NM, Beulens JW. Joint Association of Low Vitamin D and Vitamin K Status With Blood Pressure and Hypertension. Hypertension. 2017 Jun;69(6):1165-1172. doi: 10.1161/HYPERTENSIONAHA.116.08869. Epub 2017 Apr 10. PMID 28396533
- [Background] Akoko BM, Fon PN, Ngu RC, Ngu KB. Knowledge of Hypertension and Compliance with Therapy Among Hypertensive Patients in the Bamenda Health District of Cameroon: A Cross-sectional Study. Cardiol Ther. 2017 Jun;6(1):53-67. doi: 10.1007/s40119-016-0079-x. Epub 2016 Dec 29. PMID 28035630
- [Background] Nagai Y, Nakanishi K, Yamanaka N. Direct Renin Inhibitor is Better than Angiotensin II Receptor Blocker for Intrarenal Arterioles. Kidney Blood Press Res. 2016;41(5):561-569. doi: 10.1159/000443459. Epub 2016 Aug 24. PMID 27553090
- [Background] Lauro M, Carbone C, Auditore R, Musumeci T, Santagati N, Aquino R, et al. A new inclusion complex of amlodipine besylate and soluble β-cyclodextrin polymer preparation, characterization and dissolution profile. Journal of Inclusion Phenomena and Macrocyclic Chemistry. 2013;76(1-2)19-28.